CLINICAL TRIAL: NCT03146221
Title: Search for Restenosis Markers in Lower Limb Arteritis
Acronym: FEMIA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator wish
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0004
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Restenosis; Lower Limb Arteritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Person to be surgically treated for arteritis (Other)
  Interventions: Other: To look for serum microRNA profiles associated with restenosis

INTERVENTIONS:
Other: To look for serum microRNA profiles associated with restenosis — To look for serum microRNA profiles associated with restenosis

SUMMARY:
The initial hypothesis of this work is that the genesis and the evolution of the atheromatous plaque are partly controlled at the molecular level and in particular by the microRNAs through their role as regulator of the genes.

The study of the tissue and serum profile over time of specific microRNAs involved in the regulation of atheromatous plaque correlated with clinical data and restenosis imaging will allow to define biological markers of restenosis in the patient with an arteritis of the lower limbs .

This study is a pioneer in the field and it would be imprudent to conclude that a biomarker would be used clinically at the end of this work alone. Nevertheless this study will make a major advance in this topic, in vivo intervention studies with inhibition or over-expression of microRNA will obviously be necessary to confirm the use of these as biomarkers of arteritis of the lower limbs.

Regular assay of reliable biomarkers in arterial patients will ultimately suggest early management to best adapt surgical and medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any person to be surgically treated for arteritis on the femoropoplitetic stage,
* affiliated to a social security scheme,
* informed of the study and not opposed to it.

Exclusion Criteria:

* Any person taken in charge for an arteritis on the femoro-popliteal floor refusing to participate in the study,
* or not being able to express its consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-20 (Estimated); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Study of the tissue and serum profile of microRNAs by quantification by real-time PCR | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France